CLINICAL TRIAL: NCT04086394
Title: Use of PECS Block in Partial Mastectomy for Postoperative Pain Control and Mitigation of Narcotic Use- A Randomized Control Trial
Brief Title: PECS Block in Partial Mastectomy for Postoperative Pain Control
Acronym: PECS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Main Line Health (Other)
Responsible Party: Principal Investigator, Kaitlyn Kennard MD, Post Doctoral Research Fellow, Main Line Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R20-3896L
Record Dates: First submitted 2019-09-10; First posted 2019-09-11 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer; Postoperative Pain; Opioid Use; Local Anesthesia
Keywords: Pain; Narcotics; Nerve block
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Pain | interventions — Surgical Procedures, Operative; Nerve Block

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinded randomized control trial in which patient was unaware of treatment arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS Block (Experimental): Group who was randomly selected to receive the intraoperative nerve block.
  Interventions: Procedure: Pectoral Nerve Block
- Control (Sham Comparator): Patient who was randomly selected not to receive intraoperative nerve block
  Interventions: Procedure: Surgery without Nerve Block

INTERVENTIONS:
Procedure: Pectoral Nerve Block — Patients who were given 20 cc of 0.25% Marcaine as part of the pectoralis nerve block
  Arms: PECS Block
Procedure: Surgery without Nerve Block — Patient's underwent indicated procedure without regional pectoralis nerve block
  Arms: Control

SUMMARY:
The aim of this study is to evaluate patients who are undergoing partial mastectomy or removal of breast tissue and see if a pectoralis nerve block (PECS) can provide a meaningful improvement in postoperative pain control over standard pain medication. The hope is that this will decrease the need for postoperative narcotics. Prior studies have shown improved pain control using a PECS block in patients who undergo a mastectomy. PECS block is a procedure in which local anesthesia, similar to that used by dentists, is injected in the muscles of your chest and arm pit during your surgical procedure while you are asleep. This anesthetizes the nerves in the area which decreases pain. The local anesthetic used is called Marcaine. Marcaine is the brand name for bupivacaine hydrochloride which is an anesthetic known for its long duration in comparison to lidocaine.

It is known that postoperative pain is a risk factor for chronic pain which is tied to increased narcotic use. Due to the opioid epidemic considerable time and research has gone into decreasing opioid use particularly in post-operative period. The PECS block procedure involves injecting local anesthesia between two chest muscles called pectoralis major and pectoralis minor. There is an additional injection between the pectoralis minor and serratus anterior which is another muscle of the chest.

This study will be conducted at Lankenau Medical Center of Main Line Health. You have been selected since you will be undergoing a partial mastectomy (removal of a part of your breast). It is believed that PECS block has the potential to benefit your postoperative pain control. A total of 130 patients will be recruited and 65 will be placed into the treatment arm (receive intraoperative nerve block) and 65 will be placed into the non- treatment arm (no nerve block) for comparison.

DETAILED DESCRIPTION:
Prior investigations have shown that use of intraoperative PECS blocks in patients undergoing a Modified Radical Mastectomy improves postoperative pain control and decreases postoperative narcotic use which will eventually mitigate the issue of dependence on narcotics postoperatively (Kulhari et al, Blanco et al). The aim of this study is to do a prospective randomized control of patients undergoing a Partial Mastectomy at Lankenau Medical Center to see if pectoral nerve block (PECS) provides a meaningful improvement in postoperative pain control over standard pain medication as well as a decrease in postoperative narcotic use.

PECS block as described by Blanco et al has been used safely and effectively used for modified radical mastectomy in multiple studies as reviewed above (Blanco et al, Kumar et al, Kulhari et al). The breast surgeons at Lankenau Medical Center within Main Line Health are currently using the PECS block as part of their partial mastectomy procedure and have been since 5/1/19. The PECS block is currently being used at random when time and resources allow There are not certain subsets or patients who are selected for this procedure. This procedure has been well tolerated by patients and has proved feasible for the surgeons and surgical team to facilitate. Therefore since PECS block for partial mastectomy are within the standard of care at Lankenau Medical Center this study only introduces a risk of randomization rather than the increased risk of the procedure itself.

This is a randomized prospective control study looking at patients at Lankenau Hospital undergoing partial mastectomy from 8/30/19- 8/30/20 after obtaining Institutional Review Board (IRB) approval. The plan is to recruit 130 patients with 65 patients randomized into each cohort. One cohort will receive the PECS II block intraoperatively and one cohort will not. This will be a single blinded randomized control trial in that the surgeon knows who will be receiving the block however the patient will be blinded. Patient must be able to provide their own consent to be included in this study. There will be no advertisement or compensation for this study. The study will be explained to the eligible candidates at time of discussion of their surgery. Patients will be informed that involvement in the study does not affect their ability to seek or receive care at this facility.

A written informed consent will be obtained from all patients. The patients once scheduled for surgery unit will be enrolled in research study by an independent research assistant. The participants will be allocated randomly into two groups according to block randomization schedule shown below. Group one will receive anesthesia only and Group two will receive anesthesia and PECS block. The surgeon who will be performing the intraoperative block will be informed of the random and independent assignment prior to surgery. The patients will be instructed on usage of a 10-mm Visual Analogue Scale (VAS) for pain graded from 0 (no pain) to 10 (most severe pain) before surgery. Patients will be blinded as to whether or not they will be receiving intraoperative PECS block. In both the control and test groups, patients will receive general anesthesia with laryngeal mask airway or endotracheal tube per anesthesiologist discretion. Induction of anesthesia will use fentanyl 1 μg/kg and propofol 1.5-2 mg/kg until loss of verbal response with or without muscle relaxant as needed. Maintenance of anesthesia will be assessed for any intraoperative rise in heart rate and systolic blood pressure more than 20% from pre-induction value. If this occurs fentanyl 0.25 μg/kg can be administered IV. Toradol should be given unless contraindication at the end of the case. No ketamine or dilaudid will be used. Long acting opioids will be avoided. Once anesthesia is instituted prior to prepping and draping a timeout will be called during which patient will be identified and procedures to be performed will be identified.

Procedures The patient will be kept in supine position with ipsilateral arm in abducted position. The skin overlying the ipsilateral breast and adjoining infraclavicular and axillary regions will be disinfected with chloraprep and sterile draping of the area is performed. A linear ultrasound probe of high frequency (6-13 MHz) of a portable ultrasound system (Sonosite, Micromaxx Bothell, Washington USA) is taken. The probe will be covered with a sterile transparent dressing and a sterile conductivity gel will be applied. The imaging depth on the ultrasound screen is set to 4-6 cm. The ultrasound probe will first be placed cephalocaudally in the infraclavicular region and moved laterally to locate vessels directly above the 1st rib. With further lateral and downward movements the 3rd and 4th ribs will be identified. The probe is maneuvered and appropriate anatomical structures including pectoralis major and minor muscles and serratus anterior muscle are identified.

The interface between pectoralis major, pectoralis minor and serratus anterior are identified. A spinal needle 20 gauge and 4 inches in length will be used to instill 10 cc of 0.2% Marcaine between serratus anterior and pectoralis minor. Aspiration is continuously used to confirm that there is no intravenous or intra-arterial injection of local anesthesia. The needle will then be withdrawn slightly, and 10 cc of 0.25% Marcaine is injected between pectoralis major and pectoralis minor under direct ultrasound visualization. Attention is then turned to the axilla of the operative side. A spinal needle under direct visualization is used to deliver 10 cc of 0.25% Marcaine between latissimus dorsi and serratus anterior. The PECS block is finished, and the rest of the procedure is performed according to surgeon discretion. All patients whether or not they receive the PECS block will receive 10 cc of 0.25% Marcaine subcutaneously at incision site.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are patients are undergoing a partial mastectomy or excisional biopsy. Patients may undergo additional procedures such as sentinel lymph node biopsy or axillary lymph node dissection which will be recorded.

Exclusion Criteria:

* Chronic Pain, Presence of Breast Implants prior to surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | Immediately postoperatively until day 3
  Visual Analogue Pain scores scaled from 1-10 with 1 being no pain and 10 being worst pain of one's life. This scale is used to assess postoperative pain. Scores will be compared between the two groups.

SECONDARY OUTCOMES:
Postoperative Narcotic Use | 72 hours
  Amount of pain medication in morphine equivalents used after surgery until day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Kaitlyn Kennard, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Background] Kulhari S, Bharti N, Bala I, Arora S, Singh G. Efficacy of pectoral nerve block versus thoracic paravertebral block for postoperative analgesia after radical mastectomy: a randomized controlled trial. Br J Anaesth. 2016 Sep;117(3):382-6. doi: 10.1093/bja/aew223. PMID 27543533
- [Background] Kumar S, Goel D, Sharma SK, Ahmad S, Dwivedi P, Deo N, Rani R. A randomised controlled study of the post-operative analgesic efficacy of ultrasound-guided pectoral nerve block in the first 24 h after modified radical mastectomy. Indian J Anaesth. 2018 Jun;62(6):436-442. doi: 10.4103/ija.IJA_523_17. PMID 29962525
- [Background] Zhao J, Han F, Yang Y, Li H, Li Z. Pectoral nerve block in anesthesia for modified radical mastectomy: A meta-analysis based on randomized controlled trials. Medicine (Baltimore). 2019 May;98(18):e15423. doi: 10.1097/MD.0000000000015423. PMID 31045802
- [Background] Senapathi TGA, Widnyana IMG, Aribawa IGNM, Jaya AAGPS, Junaedi IMD. Combined ultrasound-guided Pecs II block and general anesthesia are effective for reducing pain from modified radical mastectomy. J Pain Res. 2019 Apr 26;12:1353-1358. doi: 10.2147/JPR.S197669. eCollection 2019. PMID 31114311
- [Background] Versyck B, van Geffen GJ, Chin KJ. Analgesic efficacy of the Pecs II block: a systematic review and meta-analysis. Anaesthesia. 2019 May;74(5):663-673. doi: 10.1111/anae.14607. PMID 30957884